CLINICAL TRIAL: NCT01885247
Title: 4-10 Week Observational Study Comparing 3 Management Strategies for Obstructive Chronic BronchoPneumopathy (OCBP) in Common Clinical Practice
Acronym: OBALPA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: 2012-746
Record Dates: First submitted 2013-05-27; First posted 2013-06-24 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Obstructive Chronic BronchoPneumopathy (OCBP)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The management of patients with Obstructive Chronic BronchoPneumopathy (OCBP) is based on a progression of therapeutic options and on a sensitization to physical activity.

For these patients selected on OCBP stage 2, the treatment options include Long Acting Beta-Agonist Bronchodilator (LABA) or Long Acting Muscarinic Antagonist Anticholinergic (LAMA) or both (LAMA+LABA).

The purpose of this study is to observe in common clinical practice the benefit of physical activity on quality of life, dyspnoea and walking distance for these patients under treatment (LABA and/or LAMA) and to determine whether these 3 medical strategies (LABA/LAMA/LABA+LAMA) benefit from physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Obstructive Chronic BronchoPneumopathy stage ≥ 2.
* Patients under treatment with LABA or LAMA or LABA+LAMA since at least 1 month.
* VEMS/CVF<70%
* VEMS<80%
* Patients without regular physical activity and without physical activity program since 1 year.

Exclusion Criteria:

* Patients under treatment with LABA + inhaled Corticoids.
* Contraindication to physical activity.
* Patients with previous history of respiratory exacerbations.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Obstructive Chronic BronchoPneumopathy (OCBP) stage ≥ 2
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life after 4 to 10 weeks of physical activity program | Visit 1 before physical activity program and Visit 2 after 4 to 10 weeks of physical activity program
  Evaluation of quality of life by specific questionnaires (VQ11, RICCI Test) and by specific parameters such as: spirometry, dyspnea, Body Mass Index (BMI), 6 minute Stepper Test (TS6), Body mass index, airflow Obstruction, Dyspnea and Exercise tolerance (BODE), O2 maximal Volume (VO2max) or Electrocardiogram (ECG).

SECONDARY OUTCOMES:
Medical Research Council dyspnea scale (grade degree 0 to 4)activity | Grade degree of dyspnea will be evaluated one time before and after the physical activity program an expected average of 10 weeks.
  Grade Degree of breathlessness related to activities (o to 4) :
  0 : Not troubled by breathlessness except on strenuous exercise
  1. : Short of breath when hurrying or walking up a slight hill
  2. : Walks slower than contemporaries on level ground because of breathlessness, or has to stop for breath when walking at own pace
  3. : Stops for breath after walking about 100m or after a few minutes on level ground
  4. : Too breathless to leave the house, or breathless when dressing or undressing
6 Minute Walking Test (6MWT) (unit : meter) | 6MWT will be realized one time before and after the physical activity program an expected average of 10 weeks.
  The original purpose of the six minute walk was to test exercise tolerance in chronic respiratory disease and heart failure. The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes.
Actimetry by accelerometer (unit : number of body movement) | Accelerometer will be installed one time before and after the physical activity program an expected average of 10 weeks.
  Actimetry by accelerometer to assess physical activity. Technically, an accelerometer consists of a device with a piezoelectric sensor that registers physical activity via body movement (acceleration) produced during a limited period of time.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Devouassoux, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France